CLINICAL TRIAL: NCT02477111
Title: A Multicenter, Open Label, Prospective, Post Approval Study of the INCRAFT® Abdominal Aortic Aneurysm (AAA) Stent Graft System in Subjects With Abdominal Aortic Aneurysms
Brief Title: European (EU) Post Approval Study of the INCRAFT® AAA Stent Graft System in Subjects With Abdominal Aortic Aneurysms
Acronym: INSIGHT
Status: Completed | Type: Observational
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Sponsor
Other Study IDs: P13-4601
Record Dates: First submitted 2015-05-30; First posted 2015-06-22 (Estimated); Results first posted 2021-04-22 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2023-11

CONDITIONS: Abdominal Aortic Aneurysms
Keywords: Endovascular repair
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Endovascular abdominal aortic aneurysm repair — Subjects with infrarenal abdominal aortic aneurysms who meet all inclusion criteria and none of the exclusion criteria will be treated with the INCRAFT Stent Graft System.

SUMMARY:
INSIGHT is a postmarket clinical follow-up study in the European Union. The purpose of the study is to continue to evaluate the safety and effectiveness/performance of INCRAFT in subjects with abdominal aortic aneurysms requiring endovascular repair in routine clinical practice. Approximately 150 subjects will be enrolled and followed through 5-years post procedure. Up to 25 sites in Europe may participate.

DETAILED DESCRIPTION:
INSIGHT is a postmarket clinical follow-up study in the European Union. The purpose of the study is to continue to evaluate the safety and effectiveness/performance of INCRAFT in subjects with abdominal aortic aneurysms requiring endovascular repair in routine clinical practice. Approximately 150 subjects will be enrolled and followed through 5-years postprocedure. Up to 25 sites in Europe may participate. Subjects will be enrolled and followed at 1 month and 6 month post-procedure and annually up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female age 18 years or older
2. Femoral access vessels should be adequate to fit the selected delivery system
3. Proximal neck length ≥ 10mm
4. Aortic neck diameters ≥ 17mm and ≤ 31mm
5. Aortic neck suitable for suprarenal fixation
6. Infrarenal and suprarenal neck angulation ≤ 60°
7. Iliac fixation length ≥ 15mm
8. Iliac diameters ≥ 7mm and ≤ 22mm
9. Minimum overall AAA treatment length (proximal landing location to distal landing location) ≥ 128mm
10. Morphology suitable for aneurysm repair
11. Provide written informed consent and as applicable written confidentiality authorization prior to initiation of study procedures
12. Subject is willing to comply with the specified follow-up evaluation schedule

Exclusion Criteria:

1. Subject has one of the following:

   1. Aneurysm sac rupture or leaking abdominal aortic aneurysm
   2. Mycotic, dissecting, or inflammatory abdominal aortic aneurysm
2. Known allergy or intolerance to nickel titanium (nitinol), Polyethylene terephthalate (PET), or polytetrafluoroethylene (PTFE)
3. Known contraindication to undergoing angiography or anticoagulation
4. Existing AAA surgical graft and/or a AAA stent-graft system
5. Women of child bearing potential whom are pregnant, lactating, or planning to become pregnant during the course of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are eligible for endovascular repair of an abdominal aortic aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2016-10-24 (Actual); Study Completion 2021-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Torsello, MD, PhD, Principal Investigator — Universitätsklinikum Münster; Jean-Pierre Becquemin, MD, PhD, Principal Investigator — CHU Henri Mondor
Locations (23):
- France (2):
  - Hospital Universitaire de Bordeaux, Bordeaux
  - Hopital Prive Paul d'Egine, Champigny-sur-Marne
- Germany (6):
  - Augusta Krankenhaus, Düsseldorf
  - University Hospital Schleswig - Holstein, Kiel
  - University Medical Center Leipzig, Leipzig
  - Universitätsklinikum Münster, Münster
  - St.-Franziskus-Hospital, Münster
  - Universitätsklinikum Würzburg, Würzburg
- Ireland (2):
  - Galway Clinic, Galway
  - University Hospital Galway, Galway
- Italy (4):
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Istituto Scientifico H San Raffaele, Milan
  - Ospedale S. Maria della Misericordia, Perugia
  - Azienda Ospedaleria San Camillo Forlanin, Rome
- Netherlands (2):
  - Radboud UMC, Nijmegen
  - Haga ziekenhuis, The Hague
- Spain (3):
  - Hospital Clinic University of Barcelona, Barcelona
  - Hospital de Donostia, Donostia / San Sebastian
  - Complejo Universitario Hospitalario de Ourense, Ourense
- Skane University Hospital, Malmo, Sweden
- United Kingdom (3):
  - Hull Royal Infirmary, Hull
  - Imperial College Healthcare NHS Trust St Mary's Hospital, London
  - Kings College Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Torsello G, Bertoglio L, Kellersmann R, Wever JJ, van Overhagen H, Stavroulakis K. Three-Year Safety and Efficacy of the INCRAFT Endograft for Treatment of Abdominal Aortic Aneurysms: Results of the INSIGHT Study. J Endovasc Ther. 2025 Jun;32(3):766-773. doi: 10.1177/15266028231214162. Epub 2023 Nov 30. PMID 38031973
- [Derived] Torsello G, Bertoglio L, Kellersmann R, Wever JJ, van Overhagen H, Stavroulakis K; INSIGHT study collaborators. One-year results of the INSIGHT study on endovascular treatment of abdominal aortic aneurysms. J Vasc Surg. 2022 Jun;75(6):1904-1911.e3. doi: 10.1016/j.jvs.2021.12.066. Epub 2022 Jan 5. PMID 34995719

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 25 academic medical centers between 2015 and the last participant was enrolled September 15, 2016
Pre-assignment Details: Of the 154 screened patients, 150 met inclusion criteria were enrolled in the study and 4 were screen fail.
Groups:
- InCraft® - AAA Stent Graft System: Single Arm EVAR Subjects who underwent procedure for the implant of InCraft® - AAA Stent Graft System
Period: Overall Study
Arm/Group | InCraft® - AAA Stent Graft System
Started | 150
Completed | 99 (Visit compliance for the final 5-year follow-up visit)
Not Completed | 51
Not completed — Death | 28
Not completed — Withdrawal by Subject | 19
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | InCraft® - AAA Stent Graft System
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.6 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 134
Angina [Count of Participants; unit: Participants] | 14
Arrhythmia [Count of Participants; unit: Participants] | 36
Coronary artery disease [Count of Participants; unit: Participants] | 44
Myocardial infarction [Count of Participants; unit: Participants] | 27
Percutaneous transluminal coronary angioplasty and/or stent [Count of Participants; unit: Participants] | 28
Coronary artery bypass grafting [Count of Participants; unit: Participants] | 19
Hypertension [Count of Participants; unit: Participants] | 120
Congestive heart failure [Count of Participants; unit: Participants] | 11
Family history of aneurysm [Count of Participants; unit: Participants] | 8
Transient Ischemic Attack [Count of Participants; unit: Participants] | 6
Stroke [Count of Participants; unit: Participants] | 9
Carotid endarterectomy/stent [Count of Participants; unit: Participants] | 2
Peripheral arterial disease [Count of Participants; unit: Participants] | 21
Diabetes [Count of Participants; unit: Participants] | 29
Hypercholesterolemia [Count of Participants; unit: Participants] | 68
Moderate renal insufficiency [Count of Participants; unit: Participants] | 18
Erectile disfunction [Count of Participants; unit: Participants] | 22
Chronic obstructive pulmonary disease (COPD) [Count of Participants; unit: Participants] | 35
Other chronic lung disease [Count of Participants; unit: Participants] | 8
Liver disease [Count of Participants; unit: Participants] | 3
Cancer [Count of Participants; unit: Participants] | 45
History of Smoking [Count of Participants; unit: Participants] | 122
Allergies [Count of Participants; unit: Participants] | 33
Other relevant medical history [Count of Participants; unit: Participants] — Other relevant medical history include: Anemia, Aortic Arch Aneurysm, Back Pain, Blindness, Bph, Carotid Occlusion, Depression, Diverticulosis, Dystonia, Gastritis, Gerd, Hernia, Hypogastric Aneurysm, Hypothyroidism, Kidney Stone, Macular Dengeneration, Mononucleosis, Obesity, Pain, Pneumothorax, Posterior L4-L5 Decompression, Prostate Hypertrophy, Renal Artery Stenosis, Renal Insufficiency, Rheumatoid Arthritis, Sleep Apnea, Suspicion Of Intraductal Pancreatic Mucinous Neoplasia, Thrombocytopenia, Varicosis, Wegener's Granulomatosis.
  Participants | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Adverse Events (MAE) Through 30 Days
Description: MAE rate through 30 days includes Death, Stroke/CVA, Myocardial Infarction, New onset renal failure (requiring dialysis)
Time Frame: Within 30-days post-procedure
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- InCraft® - AAA Stent Graft System: This is a single arm non-randomized study.
Arm/Group | InCraft® - AAA Stent Graft System
Number analyzed (Participants) | 150
participants | 0 [0.0 to 2.4]

2. Secondary Outcome: Number of Participants With Major Adverse Events Through 5 Years Post-Procedure
Description: MAE rate through 5 year includes Death, Stroke/CVA, Myocardial Infarction, New onset renal failure (requiring dialysis)
Time Frame: Through 5 years post-procedure
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | InCraft® - AAA Stent Graft System
Number analyzed (Participants) | 124
participants | 44 [33.604 to 55.304]

3. Secondary Outcome: Number of Participants With Technical Success at Conclusion of Index Procedure
Description: successful insertion of the delivery system through the vasculature and successful deployment of the device at the intended location
Time Frame: At the conclusion of the index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | InCraft® - AAA Stent Graft System
Number analyzed (Participants) | 150
Participants | 149

4. Secondary Outcome: Absence of Type I or III Endoleak
Description: defined as absence of type I or III endoleaks and absence of aneurysm enlargement (growth >5mm compared to the 1-month size measurement) within 1-year post-procedure as assessed by the core lab
Time Frame: Within 1 year post-procedure
Population: population analyzed only includes those that are eligible
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | InCraft® - AAA Stent Graft System
Number analyzed (Participants) | 115
participants | 108 [101.085 to 112.125]

5. Secondary Outcome: InCraft® - AAA Stent Graft System
Description: Single Arm EVAR Subjects who underwent procedure for the implant of InCraft® - AAA Stent Graft System
Time Frame: Assessed at 1 year
Population: population analyzed only includes those that are eligible
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- Absence of Stent-graft Migration (>10 mm) Assessed at 1-year: Absence of stent-graft migration (>10 mm) assessed at 1-year compared to the 1-month size measurement as confirmed by contrast CT-scan or other imaging.
Arm/Group | Absence of Stent-graft Migration (>10 mm) Assessed at 1-year
Number analyzed (Participants) | 122
participants | 122 [118.4 to 122]

6. Secondary Outcome: Number of Participants With Absence of Stent Graft Fracture Within 30-days and 1-year Post-procedure
Time Frame: Assessed within 30-days and 1-year post-procedure
Population: Core lab reported outcome based on received and readable imaging
Measure: Count of Participants; unit: Participants
Arm/Group | InCraft® - AAA Stent Graft System
Number analyzed (Participants) | 141
Participants | 141

7. Secondary Outcome: Absence of Aneurysm Sac Rupture
Time Frame: Within 1-year post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Absence of Stent-graft Migration (>10 mm) Assessed at 1-year
Number analyzed (Participants) | 138
Participants | 138

8. Secondary Outcome: Duration of INCRAFT® Procedure (Minutes)
Description: Duration of INCRAFT procedure is from bifurcate insertion to completion of angiography
Time Frame: Duration of INCRAFT procedure is from bifurcate insertion to completion of angiography
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | InCraft® - AAA Stent Graft System
Number analyzed (Participants) | 150
minutes | 42.3 [39.4 to 45.2]

9. Secondary Outcome: Amount of Time Fluoroscopy is Used During the Procedure
Time Frame: Duration of INCRAFT procedure is from bifurcate insertion to completion of angiography
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | InCraft® - AAA Stent Graft System
Number analyzed (Participants) | 150
minutes | 17.3 [15.9 to 18.8]

10. Secondary Outcome: Amount of Contrast Volume Used During the Procedure
Time Frame: Duration of INCRAFT procedure is from bifurcate insertion to completion of angiography
Measure: Mean (95% Confidence Interval); unit: ml
Arm/Group | InCraft® - AAA Stent Graft System
Number analyzed (Participants) | 150
ml | 99.4 [92.0 to 106.7]

ADVERSE EVENTS:
Time Frame: Adverse events are collected from index procedure until completion of study or early termination
Description: All-cause mortality, Serious Adverse Events, other (Not including serious) Adverse Events
Groups:
- INSIGHT: Single Arm EVAR Subjects who underwent procedure for the implant of InCraft® - AAA Stent Graft System
Arm/Group | INSIGHT
All-Cause Mortality (participants affected / at risk) | 28/124
Serious Adverse Events (participants affected / at risk) | 21/104
Other Adverse Events (participants affected / at risk) | 22/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | INSIGHT (N=104)
Cardiac disorders (Cardiac disorders) | 5
Gastrointestinal disorders (Gastrointestinal disorders) | 3
General disorders and administration site conditions (General disorders) | 0
Immune system disorders (Immune system disorders) | 0
Infections and infestations (Infections and infestations) | 5
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 0
Neoplasms benign, malignant and unspecified (including cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nervous system disorders (Nervous system disorders) | 3
Renal and urinary disorders (Renal and urinary disorders) | 0
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1
Surgical and medical procedures (Surgical and medical procedures) | 0
Vascular disorders (Vascular disorders) | 2
Hepatobiliary disorders (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | INSIGHT (N=104)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1
Cardiac arrhythmias (Cardiac disorders) | 1
General disorders and administration site conditions (General disorders) | 5
Infections and infestations (Infections and infestations) | 3
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0
Investigations (Investigations) | 0
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1
Nervous system disorders (Nervous system disorders) | 0
Product issues (Product Issues) | 0
Psychiatric disorders (Psychiatric disorders) | 0
Renal and urinary disorders (Renal and urinary disorders) | 1
Reproductive system and breast disorders (Reproductive system and breast disorders) | 0
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1
Surgical and medical procedures (Surgical and medical procedures) | 0
Vascular disorders (Vascular disorders) | 7
Congenital, familial and genetic disorders (Congenital, familial and genetic disorders) | 1
Eye disorders (Eye disorders) | 1
Gastrointestinal disorders (Gastrointestinal disorders) | 4
Hepatobiliary disorders (Hepatobiliary disorders) | 1
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1
Neoplasms benign, malignant and unspecified (including cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

LIMITATIONS AND CAVEATS:
Number of participants at risk my vary depending on varying windows used for analysis, imaging availability, visits completed and will therefore not be consistent throughout report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes